CLINICAL TRIAL: NCT02038283
Title: A Study on Health-related Quality of Life of Patients With Colorectal Neoplasm and Cost-Effectiveness Analysis of Colorectal Cancer Screening in Hong Kong
Brief Title: Quality of Life of Patients With Colorectal Neoplasm and Cost-Effectiveness Analysis of Colorectal Cancer Screening
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Head and Clinical Professor, The University of Hong Kong
Other Study IDs: HKCTR-973
Record Dates: First submitted 2013-08-28; First posted 2014-01-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Early Detection of Cancer; Quality of Life; Quality-Adjusted Life Years; Direct Service Costs; Cost-Benefit Analysis
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Low-risk Colorectal Polyps: ≤2 adenomas or 3-4 adenomas all of which are <1cm
- High-risk Colorectal Polyps: ≥5 adenomas or ≥3 adenomas at least one of which is ≥1cm
- Stage I CRC: at least six months since diagnosis of Stage I CRC
- Stage II CRC: at least six months since diagnosis of Stage II CRC
- Stage III CRC: at least six months since diagnosis of Stage III CRC
- Stage IV CRC: at least six months since diagnosis of Stage IV CRC

SUMMARY:
Introduction: Colorectal cancer (CRC) is the second most common cancer among Chinese in Hong Kong and the second leading cause of cancer death in this population. Several screening strategies has been associated with improved survival and may affect patients' health-related quality of life (HRQOL). HRQOL impact should be used to adjust for survival in terms of quality adjusted life years (QALY) in the evaluation of cost-effectiveness of any intervention including screening.

Objectives: to determine the HRQOL and health preference of patients with different stages of colorectal neoplasm, and to determine the most cost-effective CRC screening strategy for increasing QALYs.

Design and Subjects: A longitudinal survey to collect data on HRQOL associated with colorectal neoplasm for Markov modeling on cost-effectiveness of CRC screening. A stratified sample of 420 patients with colorectal polyps and different stages of CRC will be recruited from colorectal clinics of Queen Mary Hospital for health preference and HRQOL assessment. The HRQOL over time will be measured at baseline, 6 and 12 months later. Health preference data will be integrated with cost and effectiveness data obtained from the literature to determine the cost-effectiveness of currently recommended CRC screening strategies by Markov modeling.

Main outcome measures: The primary outcome measure is the SF-6D health preference value and QALYs. Secondary outcomes are the SF-12v2 and FACT-C scores. The outcomes will be compared between patients with different stages of colorectal neoplasm. Markov modeling study will estimate the expected QALYs gained and incremental cost-effectiveness ratio for each CRC screening strategy.

Results: The study will provide information on HRQOL of patients with colorectal neoplasm to guide health services. The Markov Model will identify the most cost-effective CRC screening strategy for Hong Kong Chinese, which can inform policy makers and the public for the prevention of CRC of the population.

DETAILED DESCRIPTION:
The aims are to determine the HRQOL and health preference (utility) of different stages of colorectal neoplasm in order to evaluate the cost-effectiveness of different CRC screening strategies for the Chinese population in Hong Kong.

The specific objectives are:

1. To determine the HRQOL preference values of patients in different stage of colorectal neoplasm in order to estimate the quality of life adjustment applicable to each stage of colorectal neoplasm.
2. To evaluate the HRQOL of patients with colorectal neoplasm in order to find out their concerns and needs.
3. To find out whether HRQOL preference of people with colorectal neoplasm changes with time.
4. To determine the expected life years gained from the reduction in the incidence and mortality rates of CRC for each CRC screening strategy base on literature review.
5. To determine the QALY gained from each CRC strategy by combining the preference value with life years gained.
6. To identify the most cost-effective CRC screening strategy and to determine the incremental cost per additional QALY gained compared to no screening, by Markov modelling.

The study hypotheses are:

1. Patients with colorectal neoplasm including those with polyps have lower HRQOL than the general population.
2. There is a gradient reduction in HRQOL preference among patients with different stages colorectal neoplasm from polyp to metastatic cancer.
3. HRQOL preference of patients with colorectal neoplasm is stable if there is no change in the disease stage.
4. Annual I-FOBT is the most cost-effective CRC screening strategy for the Chinese population in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Have life expectancy of at least 6 months
* Have confirmed diagnosis of any of the following colorectal neoplasm classified by the screening surveillance guideline and UICC/AJCC (TNM) staging system
* Have given consent to take part in the study

Exclusion Criteria:

* Inability to understand or communicate in Cantonese or Chinese
* Significant cognitive impairment judged by the doctor to be unable to answer the questionnaire
* Too ill to carry out an interview
* Refuse to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Chinese patients of 18 years old or above with a histology of confirmed colorectal polyp or cancer for at least six months were recruited from specialist outpatient medical and surgical colorectal clinics of Queen Mary hospital in Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
SF-6D Preference-based Value | Twelve months
  HRQOL preference value measured by The Chinese (HK) SF-6D Health Survey was calculated by the HK population specific algorithm. It ranges from 0 (death) to 1 (perfect health).
Quality-adjusted life years for each screening strategy | Baseline
  The effectiveness of CRC screening is quantified by Quality-adjusted life years, which was calculated as the product of average duration of each health state (including no illness) and the SF-6D preference value for that particular health state.
Direct Health Care Costs for each CRC screening strategy | Baseline
  The direct health care costs of different CRC screening strategies and treatments of different stages of CRC were estimated using the costs published by the Government Gazette.

SECONDARY OUTCOMES:
HRQOL by SF-12v2 and FACT-C | Twelve months
  HRQOL measured by the SF-12v2 and FACT-C was evaluated to identify the major problems of life of CRC patients.
Health Service Utilizations | Baseline
  Health service utilizations of patients with colorectal neoplasm were assessed to investigate their associations with HRQOL.
Factors Associated with HRQOL | Baseline
  Factors including type of treatments that may affect HRQOL of patients with CRC were explored.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Principal Investigator — Department of Family Medicine and Primary Care, Faculty of Medicine, The University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Department of Clinical Oncology, Faculty of Medicine, The University of Hong Kong, Hong Kong Island
  - Department of Medicine, Queen Mary Hospital, Hong Kong Island
  - Department of Surgery, Faculty of Medicine, The University of Hong Kong, Hong Kong Island

REFERENCES:
- [Result] Wong CK, Lam CL, Law WL, Poon JT, Chan P, Kwong DL, Tsang J. Validity and reliability study on traditional Chinese FACT-C in Chinese patients with colorectal neoplasm. J Eval Clin Pract. 2012 Dec;18(6):1186-95. doi: 10.1111/j.1365-2753.2011.01753.x. Epub 2011 Aug 18. PMID 21851512
- [Result] Wong CK, Lam CL, Poon JT, McGhee SM, Law WL, Kwong DL, Tsang J, Chan P. Direct medical costs of care for Chinese patients with colorectal neoplasia: a health care service provider perspective. J Eval Clin Pract. 2012 Dec;18(6):1203-10. doi: 10.1111/j.1365-2753.2011.01776.x. Epub 2011 Nov 23. PMID 22111837
- [Result] Wong CK, Lam CL, Rowen D, McGhee SM, Ma KP, Law WL, Poon JT, Chan P, Kwong DL, Tsang J. Mapping the Functional Assessment of Cancer Therapy-general or -Colorectal to SF-6D in Chinese patients with colorectal neoplasm. Value Health. 2012 May;15(3):495-503. doi: 10.1016/j.jval.2011.12.009. Epub 2012 Feb 17. PMID 22583460
- [Result] Wong CK, Lam CL, Mulhern B, Law WL, Poon JT, Kwong DL, Tsang J. Measurement invariance of the Functional Assessment of Cancer Therapy-Colorectal quality-of-life instrument among modes of administration. Qual Life Res. 2013 Aug;22(6):1415-26. doi: 10.1007/s11136-012-0272-x. Epub 2012 Sep 28. PMID 23054490
- [Result] Wong CK, Lam CL, Poon JT, Kwong DL. Clinical correlates of health preference and generic health-related quality of life in patients with colorectal neoplasms. PLoS One. 2013;8(3):e58341. doi: 10.1371/journal.pone.0058341. Epub 2013 Mar 13. PMID 23516465
- [Result] Wong CK, Lam CL, Law WL, Poon JT, Kwong DL, Tsang J, Wan YF. Condition-specific measure was more responsive than generic measure in colorectal cancer: all but social domains. J Clin Epidemiol. 2013 May;66(5):557-65. doi: 10.1016/j.jclinepi.2012.11.010. Epub 2013 Feb 8. PMID 23548135
- [Result] Wong CK, Lam CL, Wan YF, Rowen D. Predicting SF-6D from the European Organization for Treatment and Research of Cancer Quality of Life Questionnaire scores in patients with colorectal cancer. Value Health. 2013 Mar-Apr;16(2):373-84. doi: 10.1016/j.jval.2012.12.004. PMID 23538190
- [Result] Wong CK, Mulhern B, Wan YF, Lam CL. Responsiveness was similar between direct and mapped SF-6D in colorectal cancer patients who declined. J Clin Epidemiol. 2014 Feb;67(2):219-27. doi: 10.1016/j.jclinepi.2013.08.011. Epub 2013 Nov 1. PMID 24189090
- [Result] Wong CK, Law WL, Wan YF, Poon JT, Lam CL. Health-related quality of life and risk of colorectal cancer recurrence and All-cause death among advanced stages of colorectal cancer 1-year after diagnosis. BMC Cancer. 2014 May 17;14:337. doi: 10.1186/1471-2407-14-337. PMID 24886385
- [Result] Yang Y, Wong MY, Lam CL, Wong CK. Improving the mapping of condition-specific health-related quality of life onto SF-6D score. Qual Life Res. 2014 Oct;23(8):2343-53. doi: 10.1007/s11136-014-0668-x. Epub 2014 Mar 29. PMID 24682669
- [Result] Wong CK, Chen J, Yu CL, Sham M, Lam CL. Systematic review recommends the European Organization for Research and Treatment of Cancer colorectal cancer-specific module for measuring quality of life in colorectal cancer patients. J Clin Epidemiol. 2015 Mar;68(3):266-78. doi: 10.1016/j.jclinepi.2014.09.021. Epub 2014 Nov 6. PMID 25455838
- [Result] Lam CL, Law WL, Poon JT, Chan P, Wong CK, McGhee SM, Fong DY. Health-related quality of life in patients with colorectal neoplasm and cost-effectiveness of colorectal cancer screening in Hong Kong. Hong Kong Med J. 2015 Dec;21 Suppl 6:4-8. No abstract available. PMID 26645874
- [Derived] Wong CK, Lam CL, Wan YF, Fong DY. Cost-effectiveness simulation and analysis of colorectal cancer screening in Hong Kong Chinese population: comparison amongst colonoscopy, guaiac and immunologic fecal occult blood testing. BMC Cancer. 2015 Oct 15;15:705. doi: 10.1186/s12885-015-1730-y. PMID 26471036